CLINICAL TRIAL: NCT06821022
Title: The Impact of Pain Neuroscience Education on Physical Therapy Student's Knowledge, Attitudes, Beliefs, and Behaviours Towards Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hashemite University (Other)
Responsible Party: Principal Investigator, Ahmad Muhsen, Assistant Professor, The Hashemite University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 33/1/2024/2025
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
Keywords: Pain; Physiotherapy students; Attitudes; Education; Pain Neuroscience Education (PNE); The Revised Neurophysiology of Pain Questionnaire (RNPQ); The 13-item Modified Health Care Providers Pain and Impairment Relationship Scale (HC-PAIRS); Guideline-Concordant Low Back Pain Vignette (GCLBP-V; de novo)
MeSH Terms: conditions — Pain; Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (Experimental)
  Interventions: Other: Pain Neuroscience Education
- Red Flags Education (Active Comparator)

INTERVENTIONS:
Other: Pain Neuroscience Education — The intervention group will receive a lecture of 70min duration on pain neuroscience. The objective of this educational session is to educate students that pain can be overprotective, and that nociceptive transmission can be heavily influenced by central sensitisation (sensitivity of the central nervous system) as well as the thoughts and beliefs of the individual. The session used drawings, stories and metaphors to depict the underlying neuroscience of pain, and current pain theory.
  Arms: Pain Neuroscience Education
Other: Red Flags Education — The control group received an education session of red flags. Red flags form part of routine subjective practice for therapists as a process of screening serious or potentially sinister pathologies. Sign and symptoms for such pathologies include history of cancer, systemic symptoms such as fever or unexplained weight loss, and saddle analgesia. The red flag session will not include the neuroscience of pain.

SUMMARY:
This study investigates the effect of pain neuroscience education (PNE) on pain knowledge, attitudes, beliefs and behaviors among undergraduate physiotherapy students in Jordan

DETAILED DESCRIPTION:
Physiotherapy students at the Hashemite University will be randomly assigned into either pain neuroscience education or control lectures groups. Both groups will receive a 70-min didactic group-lecture. The control group will receive education about red-flags which are special screening questions for serious pathology. The red-flags education will discuss tissue pathology and triage for back pain classification. Neurophysiology and the biopsychosocial mode will not be discussed. The intervention group will receive a PNE lecture. All primary and secondary outcome measures consist of validated questionnaires (e.g., RNPQ, HC-PAIRS) or secondary and study-specific instruments that have undergone validation testing.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapy undergraduate students at the Hashemite University

Exclusion Criteria:

* Previous formal pain education
* Enrolled in a clinical practice module

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Revised Pain Neurophysiology Questionnaire (RNPQ) | Before and immediately after and 6 months after the education session
  The 12-item RNPQ will be used to assess knowledge of pain neurophysiology. Responses are marked yes, no or undecided. One point is awarded for correct answers. Scores range from 0 to 12, with high scores indicating good knowledge.
The modified HC-PAIRS | Prior to and immediately and 6 months after the education session
  The modified HC-PAIRS (Health Care Providers' Pain and Impairment Relationship Scale will be used to measure attitudes and beliefs towards patients with chronic pain and their ability to function. This 13-item questionnaire uses a 7-point Likert scale (strongly disagree to strongly agree). Scores range from 13 to 91 with lower scores suggesting more positive attitudes.

SECONDARY OUTCOMES:
Case vignette to measure behavior (clinical recommendations). | Before and immediately and 6 months after the education session
  A case study vignette will be used to assess clinical behavior with a chronic low back pain patient. The participants will be asked to indicate, via four multiple-choice questions their recommendations about usual daily activities, work, exercise and bed rest. The number and percentage of appropriate recommendations will be recorded. This tool is developed de novo and developed for this study to assess guideline-concordant recommendations for low back pain management. The validation process, conducted prior to participant recruitment, included [expert review for content validity, confirmatory analysis, and reliability testing].

OTHER OUTCOMES:
LBP Red-Flags Knowledge Quiz (10-item) | Baseline, Post, and 6 months after lecture control session
  It is a 10-item quiz, with yes/no answers that assesses knowledge of red-flags. Scores range from 0 to 10. This questionnaire was developed within our team. This is to provide attention-matched control content and to support participant blinding to the vignette outcome. This tool is developed de novo to provide attention-matched control content and to evaluate knowledge of red-flag indicators of serious spinal pathology. This is a de novo instrument developed and face validated for this trial. The face validation process, conducted prior to participant recruitment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hashemite University, Zarqa, Zarqa Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes
After completion of the data collection, it will be analysed and then interpreted. I will provide you with the study results and recommendations upon completion.
Supporting Information: SAP
Time Frame: After being published, the dataset and/or the statistical analyses will be made available for interested researchers upon reasonable request.
Access Criteria: After being published, the dataset and/or the statistical analyses will be made available for interested researchers upon reasonable request.

REFERENCES:
- [Background] Colleary G, O'Sullivan K, Griffin D, Ryan CG, Martin DJ. Effect of pain neurophysiology education on physiotherapy students' understanding of chronic pain, clinical recommendations and attitudes towards people with chronic pain: a randomised controlled trial. Physiotherapy. 2017 Dec;103(4):423-429. doi: 10.1016/j.physio.2017.01.006. Epub 2017 Mar 22. PMID 28797666